CLINICAL TRIAL: NCT01924949
Title: An Open-Label Study of Sofosbuvir/Ledipasvir Fixed-Dose Combination for 12 Weeks in Subjects With Nosocomial Genotype 1 HCV Infection
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination in Adults With Nosocomial Genotype 1 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0125
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2015-05

CONDITIONS: Hepatitis C
Keywords: 7977; 5885; GS-7977; GS-5885; SOF; LDV; Sofosbuvir; Ledipasvir; FDC
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDV/SOF (Experimental): Participants will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — Ledipasvir (LDV)/sofosbuvir (SOF) 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
This study is to evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in adults with nosocomial genotype 1 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 18 kg/m^2.
* HCV RNA greater than or equal to 1000 IU/mL at screening.
* Documented acquisition of nosocomial genotype 1 HCV infection within 36 months from the screening visit.
* Screening laboratory values within predefined thresholds.
* Use of two effective contraception methods if female of childbearing potential or sexually active male.
* Healthy according to medical history and physical examination with the exception of HCV diagnosis.

Exclusion Criteria:

* Unstable cardiac disease including subjects with active angina pectoris and/or hospitalization for a cardiac condition within 24 weeks prior to screening.
* Prior exposure to an HCV NS5a inhibitor.
* Pregnant or nursing female.
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
* History of solid organ transplantation.
* Current or prior history of clinical hepatic decompensation.
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol.
* Known hypersensitivity to LDV, SOF, or formulation excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Stamm, MD, PhD, Study Director — Gilead Sciences
Locations (1):
- Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 29 July 2013. The last study visit occurred on 18 August 2014.
Pre-assignment Details: 8 participants were screened.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir (LDV)/sofosbuvir (SOF) 90/400 mg fixed-dose combination (FDC) tablet once daily for 12 weeks
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Groups:
- LDV/SOF 12 Weeks: LDV/SOF 90/400 mg FDC tablet once daily for 12 weeks
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 5
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 1
    CT | 3
    TT | 1
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.58)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 3
  ≥ 800,000 IU/mL | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
percentage of participants | 100.0

2. Primary Outcome: Percentage of Participants Permanently Discontinuing Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
percentage of participants
  SVR4 | 100.0
  SVR24 | 100.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
percentage of participants
  Week 1 | 60.0
  Week 4 | 100.0
  Week 8 | 100.0
  Week 12 | 100.0

5. Secondary Outcome: HCV RNA Change From Baseline
Time Frame: Baseline; Weeks 1, 4, and 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
log10 IU/mL
  Change at Week 1 | -4.36 (0.463)
  Change at Week 4 | -4.56 (0.576)
  Change at Week 8 | -4.56 (0.576)

6. Secondary Outcome: Percentage of Participants Experiencing Virologic Failure
Description: Virologic failure was defined as
  On-treatment virologic failure:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  Virologic relapse:
  * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Baseline to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 5
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 12 Weeks
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=5)
Acute myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=5)
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Pain (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years